CLINICAL TRIAL: NCT00992459
Title: A Phase 3, Randomized, Double-Blind, Cross-Over, Active-Controlled Study of the Efficacy and Safety of HPN-100, Glyceryl Tri-(4-phenylbutyrate), for the Treatment of Adults With Urea Cycle Disorders (Help UCD)
Brief Title: Efficacy and Safety of HPN-100 for the Treatment of Adults With Urea Cycle Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HPN-100-006
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Results first posted 2013-08-12 (Estimated); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Urea Cycle Disorders
Keywords: Urea Cycle Disorder (UCD); UCD; hyperammonemia; Buphenyl (NaPBA); glycerol phenylbutyrate (GPB); Sodium Phenylbutyrate (NaPBA)
MeSH Terms: conditions — Urea Cycle Disorders, Inborn; Hyperammonemia | interventions — glycerol phenylbutyrate; 4-phenylbutyric acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Buphenyl (NaPBA) /HPN 100 Placebo (Experimental): Subjects in Arm A were randomly assigned to receive NaPBA + HPN 100 placebo for 2 weeks and then crossed over to receive HPN 100 + NaPBA Placebo for 2 weeks.
  Interventions: Drug: Buphenyl (NaPBA)
- HPN-100/NaPBA Placebo (Experimental): Subjects in Arm B were randomly assigned to receive HPN-100 + NaPBA placebo for 2 weeks and then crossed over to receive NaPBA + HPN 100 placebo for 2 weeks.
  Interventions: Drug: HPN-100

INTERVENTIONS:
Drug: HPN-100 — HPN-100 is a triglyceride that has a similar mechanism of action as NaPBA. It is a liquid with minimal taste and odor. Three teaspoons of HPN-100 (~17.4mL) delivers equivalent amount of PBA in 40 tablets of NaPBA.
  Other Names: GT4P, glyceryl tri-(4-phenylbutyrate)
  Arms: HPN-100/NaPBA Placebo
Drug: Buphenyl (NaPBA) — Buphenyl (NaPBA) will be the comparator drug to HPN-100 in this study.
  Other Names: sodium phenylbutyrate
  Arms: Buphenyl (NaPBA) /HPN 100 Placebo

SUMMARY:
This was a randomized, active-controlled, double-blind, cross-over study designed to enroll subjects with UCDs who are being treated with NaPBA.

DETAILED DESCRIPTION:
This was a randomized, active-controlled, double-blind, cross-over study designed to enroll subjects with UCDs who are being treated with NaPBA. Subjects were randomly assigned to receive either HPN-100 + NaPBA placebo or NaPBA + HPN 100 placebo for 2 weeks, and then crossed over to receive the other treatment for 2 weeks. Venous ammonia was the primary outcome measure. Subjects were admitted to the clinical research unit for 24 hours of pharmacokinetic (PK) blood and urine sampling (including an overnight stay) at the end of each treatment period, by which time the study drug had reached steady state.

Subjects followed a stable diet throughout the study as prescribed by the investigator and dietician. Throughout the study, diet diaries were completed by the subject and dietary protein intake were assessed by a dietician based on completed dietary diaries and consultation with the subject.

Subjects who completed this study and met the study entry criteria, were offered the opportunity to enroll in the HPN-100 open-label safety protocol (HPN-100-007).

Study acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of UCD (Urea Cycle Disorder) involving deficiencies of Carbamyl phosphate synthetase (CPS), Ornithine transcarbamylase (OTC), or Arginosuccinate (ASS), confirmed via enzymatic, biochemical, or genetic testing
* Adult UCD subjects 18 years of age or older who are being treated with Buphenyl/Sodium phenylbuterate (NaPBA) for their UCD; subjects must be on a stable dose of NaPBA for at least 1 week prior to the Day 1 visit. Subjects who are not receiving NaPBA at the initial screening visit, but who have the potential to benefit from treatment, may start receiving NaPBA during the screening period and be enrolled as long as they are on a stable dose of NaPBA for at least 1 week prior to Day 1.
* No clinical evidence of hyperammonemia associated with an ammonia level of ≥ 100 μmol/L during the 2 weeks preceding screening
* Signed informed consent by subject
* Able to perform and comply with study activities, including blood draws and 24-hour urine samples
* Negative pregnancy test for all females of childbearing potential
* All females of childbearing age and all sexually active males must agree to use an acceptable method of contraception throughout the study. Appropriate contraceptive methods include hormonal contraceptives (oral, injected, implanted, or transdermal), tubal ligation, intrauterine device, hysterectomy, vasectomy, or double barrier methods. Abstinence is an acceptable form of birth control, though appropriate contraception must be used if the subject becomes sexually active.

Exclusion Criteria:

* Screening or baseline ammonia level of ≥ 100 μmol/L or signs and symptoms indicative of hyperammonemia during the 2-week period preceding screening or enrollment; subjects may be re-screened after their ammonia is controlled and are stable for at least 14 days, at the discretion of the investigator
* Use of any investigational drug within 30 days of Day 1
* Active infection (viral or bacterial) or any other intercurrent condition (apart from UCD) that may increase ammonia levels
* Any clinical or laboratory abnormality of Grade 3 or greater severity according to the Common Terminology Criteria for Adverse Events (CTCAE) v3.0, except Grade 3 elevations in liver enzymes, defined as levels 5-20 times upper limit of normal (ULN) in alanine aminotransferase (ALT/SGPT), aspartate aminotransferase (AST/SGOT), or gamma glutamyl transpeptidase (GGT) in a clinically stable subject
* Any clinical or laboratory abnormality or medical condition that, at the discretion of the investigator, may put the subject at increased risk by participating in this study
* Use of any medication known to significantly affect renal clearance (e.g., probenecid) or to increase protein catabolism (e.g., corticosteroids), or other medication known to increase ammonia levels (e.g., valproate), within the 24 hours prior to Day 1 and throughout the study
* Use of sodium benzoate within one week of Day 1
* History of corrected QT interval (QTc) prolongation or QTc interval > 450 msec at screening or baseline
* Known hypersensitivity to phenylacetate (PAA) or phenylbutyrate (PBA)
* Liver transplant, including hepatocellular transplant
* Breastfeeding or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (22):
- United States (21):
  - Long Beach Memorial, Long Beach, California
  - UCLA, Los Angeles, California
  - Stanford University, Stanford, California
  - Denver Children's Hospital, Aurora, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - University of Iowa, Iowa City, Iowa
  - Maine Medical Center, Portland, Maine
  - SNBL-Clinical Pharmacology Center, Baltimore, Maryland
  - Tufts-New England Medical Center, Boston, Massachusetts
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mount Sinai School of Medicine, New York, New York
  - Westchester Medical Center, Valhalla, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Diaz GA, Krivitzky LS, Mokhtarani M, Rhead W, Bartley J, Feigenbaum A, Longo N, Berquist W, Berry SA, Gallagher R, Lichter-Konecki U, Bartholomew D, Harding CO, Cederbaum S, McCandless SE, Smith W, Vockley G, Bart SA, Korson MS, Kronn D, Zori R, Merritt JL 2nd, C S Nagamani S, Mauney J, Lemons C, Dickinson K, Moors TL, Coakley DF, Scharschmidt BF, Lee B. Ammonia control and neurocognitive outcome among urea cycle disorder patients treated with glycerol phenylbutyrate. Hepatology. 2013 Jun;57(6):2171-9. doi: 10.1002/hep.26058. Epub 2013 Jan 3. PMID 22961727
- [Derived] Mokhtarani M, Diaz GA, Rhead W, Berry SA, Lichter-Konecki U, Feigenbaum A, Schulze A, Longo N, Bartley J, Berquist W, Gallagher R, Smith W, McCandless SE, Harding C, Rockey DC, Vierling JM, Mantry P, Ghabril M, Brown RS Jr, Dickinson K, Moors T, Norris C, Coakley D, Milikien DA, Nagamani SC, Lemons C, Lee B, Scharschmidt BF. Elevated phenylacetic acid levels do not correlate with adverse events in patients with urea cycle disorders or hepatic encephalopathy and can be predicted based on the plasma PAA to PAGN ratio. Mol Genet Metab. 2013 Dec;110(4):446-53. doi: 10.1016/j.ymgme.2013.09.017. Epub 2013 Oct 8. PMID 24144944

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty six subjects were screened and randomized at the participating sites between October 2009 to August 2010.
Pre-assignment Details: There were no screen failures.
Groups:
- Arm A: Subjects in Arm A were assigned to receive NaPBA + HPN 100 placebo for 2 weeks All patients in Arm A received HPN100 placebo (+ concomitant active NaPBA)
- Arm B: Subjects in Arm B were assigned to receive HPN-100 + NaPBA placebo for 2 weeks All patients in Arm B received NaPBA placebo (+ concomitant active HPN 100)
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 22 (All patients received HPN 100 placebo in Arm A (+ concomitant active NaPBA)) | 24 (All patients received NaPBA placebo in Arm B (+ concomitant active HPN 100))
Completed | 21 (Totals enrolled and completed in Arm A NaPBA treatment + HPN 100 Placebo are not mutually exclusive.) | 23 (Totals enrolled and completed in Arm B HPN 100 treatment + NaPBA Placebo are not mutually exclusive.)
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Arm A: Patients randomized to receive NaPBA + HPN 100 placebo for 2 weeks (Treatment Period 1) followed by HPN-100 + NaPBA placebo for 2 weeks (Treatment Period 2)
- Treatment Arm B: Patients randomized to receive HPN-100 + NaPBA placebo for 2 weeks (Treatment Period 1) followed by NaPBA + HPN-100 placebo for 2 weeks (Treatment Period 2)
- Total: Total of all reporting groups
Arm/Group | Treatment Arm A | Treatment Arm B | Total
Number analyzed (Participants) | 22 | 24 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 24 | 46
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32
  Male | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint Was the 24-hour Area Under the Curve for Blood Ammonia (NH324-hour AUC) on Days 14 and 28.
Description: Blood samples were collected at pre-dose, 2, 4, 8, 12, 16, 20 and 24 hours after first dose on days 14 and 28. Arm A day 14 and Arm B day 28 data were combined as a NaPBA treatment Arm. Arm B day 14 and Arm A day 28 data were combined as a HPN-100 treatment Arm.
Time Frame: pre-dose, 2, 4, 8, 12, 16, 20 and 24 hours after first dose on days 14 and 28
Population: Intent-to-Treat (ITT) (N = 45): Patients receiving any amount of NaPBA or HPN-100 comprise the ITT population. ITT population was to be used for the primary analysis of this endpoint. One subject who withdrew from study after receiving one dose of NaPBA yielding N=44
Measure: Mean (Standard Deviation); unit: μmol∙h/L
Groups:
- NaPBA: Patients treated with NaPBA
- HPN-100: Patients treated with HPN-100
Arm/Group | NaPBA | HPN-100
Number analyzed (Participants) | 44 | 44
μmol∙h/L | 976.6 (865.9) | 865.35 (660.53)

2. Secondary Outcome: Correlation Between Urinary Phenylacetylglutamine (PAGN) Excretion Over 24 Hours (U-PAGN24-hour Excr) and Venous Ammonia - Area Under the Concentration-time Curve From Time 0 (Predose) to 24 Hours (AUC0-24)
Description: The correlation between 24-hour urinary phenylacetylglutamine (PAGN) excretion (U-PAGN24-hour Excr) and venous ammonia AUC0-24 was summarized and the correlation was tested using the Spearman rank-order correlation.
Time Frame: 28 Days
Population: Intent-to-Treat (ITT) (N = 45): Patients receiving any amount of NaPBA or HPN-100 comprise the ITT population. ITT population was to be used for the primary analysis of this secondary endpoint. One subject who withdrew from study after receiving one dose of NaPBA yielding N=44
Measure: Number; unit: correlation coefficient
Arm/Group | NaPBA | HPN-100
Number analyzed (Participants) | 44 | 44
correlation coefficient | 0.437 | 0.219

3. Secondary Outcome: Maximum Ammonia Values Observed on NaPBA Versus HPN-100
Description: Blood samples were collected at pre-dose, 2, 4, 8, 12, 16, 20 and 24 hours after first dose on days 14 and 28.
Time Frame: pre-dose, 2, 4, 8, 12, 16, 20 and 24 hours after first dose on days 14 and 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | NaPBA | HPN-100
Number analyzed (Participants) | 44 | 44
µmol/L | 70.83 (66.705) | 60.94 (46.213)

4. Secondary Outcome: Rate (Percentage) of Ammonia Values Above Upper Limit of Normal (ULN) on NaPBA Versus HPN-100
Description: NaPBA treated arm: total 345 blood samples were collected. HPN-100 treated arm: 343 blood samples were collected.
Time Frame: on Day 14 and Day 28
Population: as for outcome 2
Measure: Number; unit: samples
Units Other Than Participants: blood samples
Arm/Group | NaPBA | HPN-100
Number analyzed (Participants) | 44 | 44
Number analyzed (blood samples) | 345 | 343
samples | 125 | 122

5. Secondary Outcome: Number and Severity of Symptomatic Hyperammonemic Crises
Description: Severity of symptomatic hyperammonemic crises was measured by peak ammonia level (µmol/L) when it is >= 100 µmol/L.
Time Frame: 29 Days
Population: Safety population: (N=45 for NaPBA; N = 44 for HPN): Patients receiving any amount of NaPBA or HPN-100 comprise the Safety population. Safety population was to be used for safety analysis performed.
Measure: Number; unit: events
Arm/Group | NaPBA | HPN-100
Number analyzed (Participants) | 45 | 44
events | 1 | 0

6. Secondary Outcome: Rate of Adverse Events in Each Treatment Group
Time Frame: 29 Days
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | NaPBA | HPN-100
Number analyzed (Participants) | 45 | 44
participants | 23 | 27

7. Secondary Outcome: Cmax for PAA of NaPBA and HPN-100 in Plasma
Description: Blood samples were collected at pre-dose, 2, 4, 8, 12, 16, 20 and 24 hours after first dose on days 14 and 28.
Time Frame: pre-dose, 2, 4, 8, 12, 16, 20 and 24 hours after first dose on days 14 and 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | NaPBA | HPN-100
Number analyzed (Participants) | 44 | 44
μg/mL | 52.2 (41.86) | 38.5 (39.5)

8. Secondary Outcome: Cmax for PBA of NaPBA and HPN-100 in Plasma
Description: Blood samples were collected at pre-dose, 2, 4, 8, 12, 16, 20 and 24 hours after first dose on days 14 and 28.
Time Frame: pre-dose, 2, 4, 8, 12, 16, 20 and 24 hours after first dose on days 14 and 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | NaPBA | HPN-100
Number analyzed (Participants) | 44 | 44
μg/mL | 80.9 (52.5) | 51.9 (34.87)

9. Secondary Outcome: Cmax PAGN of NaPBA and HPN-100 in Plasma
Description: Blood samples were collected at pre-dose, 2, 4, 8, 12, 16, 20 and 24 hours after first dose on days 14 and 28.
Time Frame: pre-dose, 2, 4, 8, 12, 16, 20 and 24 hours after first dose on days 14 and 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | NaPBA | HPN-100
Number analyzed (Participants) | 44 | 44
μg/mL | 78.6 (43.86) | 86.8 (44.7)

10. Secondary Outcome: U-PAGN24-hour Excr of NaPBA and HPN-100
Time Frame: 24 hours on Day 14 of each treatments
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: μg
Arm/Group | NaPBA | HPN-100
Number analyzed (Participants) | 44 | 44
μg | 13627515 (7086307.8) | 13502745 (7088941.1)

ADVERSE EVENTS:
Time Frame: 29 days
Groups:
- NaPBA: Patients received NaPBA
- HPN-100: Patients received HPN-100
Arm/Group | NaPBA | HPN-100
Serious Adverse Events (participants affected / at risk) | 1/45 | 1/44
Other Adverse Events (participants affected / at risk) | 23/45 | 27/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NaPBA (N=45) | HPN-100 (N=44)
Gastroenteritis (Infections and infestations) | 0 | 1
Hyperammonaemia (Metabolism and nutrition disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4.4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NaPBA (N=45) | HPN-100 (N=44)
Abdominal discomfort (Gastrointestinal disorders) | 3 | 0
Oral discomfort (General disorders) | 2 | 0
abdominal pain (Gastrointestinal disorders) | 2 | 3
decreased appetite (Metabolism and nutrition disorders) | 2 | 3
diarrhea (Gastrointestinal disorders) | 3 | 7
dyspepsia (General disorders) | 3 | 2
fatigue (General disorders) | 1 | 3
flatulence (Gastrointestinal disorders) | 1 | 6
food aversion (General disorders) | 2 | 1
headache (Nervous system disorders) | 4 | 6
increased appetite (Metabolism and nutrition disorders) | 2 | 0
nausea (Gastrointestinal disorders) | 3 | 1
vomiting (Gastrointestinal disorders) | 2 | 3
dizziness (Nervous system disorders) | 4 | 0
ammonia increased (Investigations) | 1 | 2
dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days